CLINICAL TRIAL: NCT07357870
Title: Safety and Effectiveness of CGB-600 Gel for the Treatment of Non-Segmental Facial Vitiligo: A Randomized, Double-Blind, Vehicle-Controlled Phase 1 Proof of Concept Study (Study No. CGB-600-02)
Brief Title: A Proof of Concept, Phase 1 Study of CGB-600 for the Topical Treatment of Non-Segmented Facial Vitiligo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGB-600-02
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGB-600 gel (Experimental)
  Interventions: Drug: Drug: CGB-600 gel, experimental drug
- vehicle gel (Placebo Comparator)
  Interventions: Other: placebo: gel vehicle

INTERVENTIONS:
Drug: Drug: CGB-600 gel, experimental drug — experimental drug
  Arms: CGB-600 gel
Other: placebo: gel vehicle — placebo gel
  Arms: vehicle gel

SUMMARY:
The goal of this clinical trial is to learn if drug CGB-600 works to treat vitiligo on the face and neck in participants between 18-60 years of age. It will also learn about the safety of CGB-600. The main questions it aims to answer are:

Does CGB-600 decrease the severity of vitiligo on the face and neck? What medical problems do participants have when taking drug CGB-600? Researchers will compare CGB-600 to a non-active drug (vehicle) to see if CGB-600 works to treat vitiligo.

Participants will:

Apply face twice daily for a period of 24 weeks. Visit the clinic 8 times for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 to 60 years old) diagnosed with non-segmental vitiligo on the face or neck. Dermoscopy and a Wood's Lamp Examination should be performed to confirm the diagnosis.
2. Facial and/or neck involvement with 1-3 vitiligo lesions (total combined area of lesions ≥ 6 cm² and ≤ 40 cm² and ≥75% depigmentation) for at least 3 months (90 days) prior to Baseline.
3. Vitiligo involvement ≤ 20% total body surface area (BSA).
4. Is otherwise in good health and free from any disease, condition, or constraint that, in the Investigator's opinion, might interfere with the conduct of the study
5. Stable disease, as judged by the investigator and patient report. Facial lesions must have been present ≤ 5 years with no new lesions or progression within 90 days prior to Baseline
6. Is not currently taking any medication for vitiligo in oral, topical, or any other form, including over-the-counter (OTC) and/or cosmetic products
7. Agrees to refrain from any other treatment modalities, including lights, lasers, or other medical devices, prescription or otherwise, for vitiligo for 4 weeks (28 days) before and during the study treatment (see Table 5.1 for complete list)
8. Agrees to refrain from using any lotions, creams, liquids, or other topical products at the treatment site during the study treatment period unless directed to do so by the investigator
9. Agrees to review and sign a written informed consent form
10. Can understand and comply with the study requirements as judged by the investigator
11. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test and must agree to use a highly effective form of contraception or abstinence and be willing to remain on that same method of birth control throughout the study.

    -

Exclusion Criteria:

* 1. Females who are pregnant, breastfeeding, or of childbearing potential and not practicing reliable birth control

  2. History of segmental or mixed vitiligo

  3. Vitiligo affecting only external genitalia or hands/feet

  4. History of skin cancer or pre-cancerous lesions in the treatment area

  5. Past use of topical or systemic vitiligo treatments within 4 weeks (28 days) prior to Baseline 6. Current active use of topical corticosteroids on the face or immunomodulatory therapies within 4 weeks (28 days) prior to Baseline

  7. Use of biological, investigational, or experimental therapy 3 months before Baseline that could potentially interfere with the study participation or assessment

  8. Known hypersensitivity to any components of the intervention or vehicle

  9. History of melanocyte-keratinocyte transplantation procedure (MKTP) or other surgical treatments for vitiligo

  10. Uncontrolled thyroid function or other medical conditions that could interfere with study participation or assessment

  11. Use within 4 weeks (28 days) prior to Baseline (washout period) of 1) oral, intravenous or intralesional corticosteroids, 2) UVA/UVB therapy, 3) non-prescription UV light sources, 4) any oral or topical Janus kinase inhibitor (JAKi), or 5) cytotoxic drugs

  12. Has demonstrated resistance to previous JAKi treatment, topical or systemic

  13. Has clinically significant laboratory anomalies or vital signs, as judged by the investigator, that would interfere with the conduct or interpretation of study results

  14. Has any inflammations or any active skin diseases on the face and/or neck including complete leukotrichia or facial lesions that would interfere with study participation or assessment

  15. Is currently participating in another investigational medication or device study or has participated in a clinical trial within 30 days of the intended start of study treatment

  16. Is unable or unwilling to comply with any of the study requirements

  17. Has medical or psychiatric conditions or a personal situation that may increase the risk associated with study participation or may interfere with interpretation of study results or subject compliance and, in the opinion of the Principal Investigator (PI), makes the subject inappropriate for study entry

  18. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Overall Incidence of tabulated safety events. [Time Frame: From enrollment to end of study at 24 weeks] | From enrollment to end of study at 24 weeks

SECONDARY OUTCOMES:
evaluate effectiveness Percent of participants achieving ≥ 50% reduction in Facial Vitiligo Area Scoring Index (F-VASI) score in the treated target area from baseline at Week 24 | from enrollment to end of study (24 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara T.C. Ministry of Health, Ankara, Turkey
  - Istanbul Universitesi faculty of Medicine, Istanbul, Turkey

IPD SHARING:
Plan to Share IPD: No